CLINICAL TRIAL: NCT02473211
Title: Efficacy and Safety of Sofosbuvir Plus Daclatasvir in Chinese Treatment-experienced Patients With Chronic Genotype 1b HCV Infection
Brief Title: SOF Plus DCV in Treating Chinese Treatment-experienced HCV Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Humanity and Health Research Centre (Other)
Collaborators: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H&H_SOF plus DCV treatment
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Chronic Hepatitis C Infection
MeSH Terms: interventions — Sofosbuvir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SOF+DCV (Experimental): Participants will receive Sofosbuvir (SOF) 400 mg and Daclatasvir (DCV) 60 mg daily for 12 weeks.
  Interventions: Drug: Sofosbuvir; Drug: Daclatasvir

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir 400 mg tablet administered once daily
  Other Names: GS-7977
Drug: Daclatasvir — Daclatasvir 60mg tablet administered once daily
  Other Names: BMS-790052

SUMMARY:
For those chronic hepatitis C patients, who are interferon-ineligible or intolerant, there is a burning need for the development of pan-oral interferon-free regimen. The investigators examine the efficacy and safety of sofosbuvir, a NS5B nucleotide polymerase inhibitor and daclatasvir, an NS5A replication complex inhibitor in Chinese treatment-experienced cirrhosis patients with chronic G1b infection.

DETAILED DESCRIPTION:
Chinese genotype 1b HCV treatment-experienced cirrhotic patients are recruited and treated with 12 weeks sofosbuvir 400 mg daily plus daclatasvir 60 mg daily. At baseline, liver stiffness measurement (LSM) using transient elastography (FibroScan®) is used to assess liver fibrosis and the single nucleotide polymorphism ofinterferon-λ 3 (IL-28, rs12979860, C or T) and IFLN4 (ss469415590, TT or ΔG) is determined. Serial measurement of plasma HCV RNA levels are performed with the use of the COBAS TaqMan real-time assay (Roche version 2.0), at baseline, Day 2,4 and 7, week 2,4 and 12, post-treatment week 12. The primary efficacy end point is a sustained virologic response 12 weeks after the end of treatment (SVR12).

ELIGIBILITY:
Inclusion Criteria:

1. Patients chronically infected with HCV Genotype-1b;
2. Documented evidence of relapse after completion of previous course of interferon-based regimen with or without ribavirin;
3. HCV RNA level greater than 10,000 IU/ml at screening;
4. Patients with compensated cirrhosis are permitted.

Exclusion Criteria:

1. Current or prior history: Clinically-significant illness (other than HCV) or any other major medical disorder that may interfere with treatment, assessment or compliance with the protocol; individuals currently under evaluation for a potentially clinically-significant illness (other than HCV) are also excluded;
2. Screening ECG with clinically significant abnormalities;
3. Laboratory results outside of acceptable ranges at screening;
4. Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with sustained virologic response 12 weeks after the end of treatment (SVR12) | Post treatment Week 12
  SVR12 is defined as HCV RNA < the lower limit of quantitation (LLOQ) (15 IU/ml) 12 weeks following the last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: George KK Lau, MD, Principal Investigator — Humanity and Health GI and Liver Centre
Locations (2):
- China (2):
  - Liver Fibrosis Diagnosis and Treatment Centre, 302 Hospital, Beijing, Beijing Municipality
  - Humanity and Health GI and Liver Centre, Hong Kong, Hong Kong